CLINICAL TRIAL: NCT04125329
Title: Umbilical Cord Mesenchymal Stem Cells Therapy for Diabetic Nephropathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43136152-9
Record Dates: First submitted 2019-09-16; First posted 2019-10-14 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Mesenchymal Stem Cells; Diabetic Nephropathy
Keywords: Human umbilical cord mesenchymal stem cells; Diabetic nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human umbilical cord mesenchymal stem cells (Experimental): Human umbilical cord mesenchymal stem cells were given to each diabetic nephropathy subject once a month, peripheral intravenous injection, a total of three times
  Interventions: Drug: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Drug: Human umbilical cord mesenchymal stem cells — Human umbilical cord mesenchymal stem cells were given to each diabetic nephropathy subject once a month, peripheral intravenous injection, a total of three times

SUMMARY:
This clinical trial assessed the safety of human umbilical cord mesenchymal stem cell therapy in 15 patients with diabetic nephropathy. Fifteen subjects received umbilical cord mesenchymal stem cell therapy 3 times. Approximately 1 × 106/kg of human umbilical cord mesenchymal stem cells were administered by peripheral intravenous infusion once a month .Endpoints:Primary endpoint: Safety and adverse events (safety and tolerability of umbilical cord mesenchymal stem cell therapy within 60 weeks).Secondary endpoint indicators:Efficacy measures: eGFR, urinary albumin-to-creatinine ratio, and percentage changes of 24-h urinary protein quantities from baseline to 60 weeks.

DETAILED DESCRIPTION:
Dosage and administration method: Fifteen subjects received umbilical cord mesenchymal stem cell therapy 3 times. Approximately 1 × 106/kg of human umbilical cord mesenchymal stem cells were administered by peripheral intravenous infusion once a month at 0, 4, and 8 weeks. Routine medications were used.

Follow-up: Patient follow-up was performed 7 times at 0, 4, 8, 20, 32, 48, and 60 weeks. Blood and urine were collected for determination of urinary albumin-to-creatinine ratio, 24-h urine protein ratio, liver and kidney function, fasting blood glucose, 2-h postprandial blood glucose, glycosylated hemoglobin, eGFR, blood lipids, and blood electrolytes at each follow-up visit. The daily dose of insulin was recorded. Blood samples were taken after each infusion of stem cells for flow cytometry and for the detection of CD3, CD4, CD8, CD28+, Treg, CD80, CD86, HLA-DR, CD83, and CD1a cells. Plasma levels of the cytokines IFN-gamma, TNF, IL-2, IL-4, IL-10, IL-6, IL-12P70, IL-8, and IL-1 beta were also determined.

Endpoints:

Primary endpoint: Safety and adverse events (safety and tolerability of umbilical cord mesenchymal stem cell therapy within 60 weeks): The number and severity of adverse events, an evaluation of their association with the umbilical cord mesenchymal stem cell treatment, and the outcome of the adverse events.

The patients' discomfort and clinical symptoms during the study period were recorded.

The subjects' relevant laboratory test indices, 12-lead electrocardiogram, vital signs, and physical examination results were recorded during the study.

Secondary endpoint indicators:

Efficacy measures: eGFR, urinary albumin-to-creatinine ratio, and percentage changes of 24-h urinary protein quantities from baseline to 60 weeks.

Data analysis:

The number of adverse events and the number of severity adverse events were determined based on the changes in the data summary (i.e., descriptive statistics).

A multilevel statistical analysis model (mixed effects model) was used to infer the relationship between treatment factors and key indicators, reflect the changing trend of key indicators in different time periods, and draw statistical analysis conclusions.

ELIGIBILITY:
Enrollment criteria:

* Adult patients (age 18-60 years) who met the WHO 1999 diagnostic criteria for type 2 diabetes, regardless of gender;
* Concomitant proteinuria ,3500 mg/day≥24h urinary protein excretion ≥500 mg/day, and uncontrolled disease course;
* Pathological examination of puncture biopsy resulting in diagnosis of type IIa, IIb, III, or IV diabetic nephropathy. (In 2010, an international expert group led by Bruijn of Leiden University in the Netherlands published a pathological classification system for diabetic nephropathy);
* eGFR between 30 ml/min/1.732 m2 and 60 ml/min/1.732 m2;
* Diabetes treatment according to guidelines and norms before the umbilical cord mesenchymal stem cell therapy;
* If there is a possibility of pregnancy in female, must be negative pregnancy test, not in lactation, and confirm that is receiving the method of contraception recognized by the researchers, and agree to maintain the method of contraception throughout the study. Sexually active male patients must agree to the use of an appropriate contraceptive method for birth control from the first administration of the study treatment until 24 weeks after the last administration.
* participate in all visits, examinations, and treatments as required by the experimental protocol.

Exclusion criteria:

* Patients with kidney biopsy diagnosis of type I diabetic nephropathy or a diagnosis of another glomerular disease;
* Patients with abnormal renal function (serum creatinine ≥ the upper limit of normal);
* Patients with HbA1c ≥10%;
* Patients with active liver disease or abnormal liver function test results (ALT or AST ≥2 times the upper limit of normal);
* Patients with blood leukocyte count <3.0 × 109/L, hemoglobin <90 g/L, platelet count <100 × 109/L, or those who have other hematologic diseases (severe anemia, idiopathic thrombocytopenic purpura, splenomegaly, coagulation dysfunction, etc.);
* Patients with serious and unstable cardiovascular or cerebrovascular diseases (unstable angina pectoris, coronary artery disease, cerebrovascular disease, transient ischemic attack, congestive heart failure, etc.), acute and difficult to control the disease, after treatment has not been effectively controlled severe hypertension (blood pressure >160/100 mm Hg), or organ transplantation;
* Patients with increased use of hypotensive drugs in the past 3 months;
* Patients with uncontrolled infection;
* Patients with tumors or abnormal tumor marker levels;
* Patients with blood-borne diseases (i.e., HIV, syphilis, hepatitis B, and hepatitis C);
* Pregnancy, the potential for pregnancy, or lactation;
* Patients receiving immunosuppressive therapy;
* Patients with a history of allergy, especially patients allergic to human blood albumin;
* Patients with mental illness affecting their voluntarism, ability to make decisions, and ability to communicate；
* A history of alcoholism or known drug addiction in the last 2 years;
* Participation in another clinical trial within the last 3 months;
* Patients judged inappropriate for this study by the physicians.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent and Treatment-Chronic Adverse Events of human umbilical cord mesenchymal stem cells for diabetic nephropathy patient | 60 weeks
  The patient's discomfort and clinical symptoms during the study were recorded, as well as the related laboratory test indicators and physical examination abnormalities of the subjects during the study.Describe the association with umbilical cord mesenchymal stem cell therapy and calculate the incidence of treatment-related acute and chronic adverse events.

SECONDARY OUTCOMES:
Changes in eGFR before and after treatment; Changes in 24h urine protein quantification before and after treatment | 60Weeks,but the major evaluated time is 12 weeks after the last treatment, compared with baseline (0W)
  Main evaluation index of curative effect:percentage changes in estimated glomerular filtration rate (eGFR), urinary albumin creatinine ratio, and 24-hour urinary protein quantification from baseline to 60 weeks of treatment. Other efficacy indicators included fasting blood glucose, blood glucose 2 hours after breakfast, HbA1c, blood and urine routine, liver and renal function, blood lipid, blood electrolyte, and daily insulin dosage.

CONTACTS AND LOCATIONS:
Locations (1):
- Yan'an Hospital of Kunming City, Kunming, China

IPD SHARING:
Plan to Share IPD: No